CLINICAL TRIAL: NCT06115434
Title: Salvage Cystectomy vs Radical Cystectomy, a Comparative Study
Brief Title: Comparing Operative, Postoperative and Quality of Life of Patients After Salvage and Radical Cystectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Salah Abdul Mawgoud, principal ivestigator, urology resident, Assiut University
Other Study IDs: Salvage and radical cystectomy
Record Dates: First submitted 2022-11-27; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-08

CONDITIONS: Urinary Bladder Cancer
Keywords: salvage; radical
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cystectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- salvage cystectomy: patients will undergo salvage cystectomy after failure of bladder preservation protocol
  Interventions: Procedure: cystectomy
- radical cystectomy: patients who will undergo radical cystectomy without going through bladder preservation
  Interventions: Procedure: cystectomy

INTERVENTIONS:
Procedure: cystectomy — cystectomy either radical or salvage involves removal of urinary bladder together with prostate, seminal vesicles and urethra with lymph node dissection.

SUMMARY:
To compare operative difficulties, type of urinary diversion, intraoperative & postoperative complications and quality of life in patients underwent radical cystectomy and those after salvage cystectomy.

DETAILED DESCRIPTION:
Radical cystectomy is the standard treatment for muscle-invasive bladder cancer. However, in well selected patients, bladder preservation with radiotherapy and chemotherapy with maximal transurethral resection of bladder tumor (TURBT) is done. Nowadays, multiple guidelines support the use of bladder sparing therapy (BST) in the form of a trimodal therapy (TMT) as an alternative to primary RC with curative intent for selected, well-informed and compliant patients, who desire to retain their bladder. Patients usually would prefer a BST, as it is considered tolerable due to its minimal invasiveness with genuinely manageable toxicity. However, a significant proportion of patients may eventually need a salvage radical cystectomy (SV-RC) due to non-response to BST or local recurrence. Salvage cystectomy post-trimodality therapy for intravesical recurrence has an intraoperative and early complication rate comparable to primary cystectomy, Salvage cystectomy post-trimodality therapy is associated with a higher risk of overall and major late complications than primary cystectomy, Irradiated tissue presents technical and surgical challenges, as radiation can lead to an overexpression of cytokines which causes uncontrolled matrix proliferation and fibrosis These post-radiation changes lead to fixation of pelvic organs, making blunt dissection more difficult, as well as causing disruption of surgical landmarks and loss of tissue planes Another consequence of irradiated tissue is that healing is impaired and tissue is weakened, leading to the potential for wound breakdown and fistula formation.

ELIGIBILITY:
Inclusion Criteria:

* patients with muscle invasive bladder cancer ≥ cT2N0/xM0 who underwent salvage cystectomy / going for bladder preservation protocol.
* patients with muscle invasive bladder cancer underwent radical cystectomy.

Exclusion Criteria:

* Patients refusing to participate in our study.
* patients with metastatic bladder cancer

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with muscle invasive bladder cancer
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-01-30 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
intraoperative and postoperative complications of salvage and radical cystectomy. | up to 1 year (retrospective and prospective case series)
  intraoperative blood loss, quality of dissection, intestinal injury.
urinary diversion | 3 months
  type of urinary diversion whether continent or incontinent and which type of shunt.

SECONDARY OUTCOMES:
quality of life of patients postoperatively | up to 3 years
  describing quality of life in patients postoperatively and how they are able to face and adapt to the new changes and requirements postoperatively
postoperative erectile function of patients | up to 2 years
  studying the effect of radical and salvage cystectomy in patients' sexual function.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moonen LM, Horenblas S, van der Voet JC, Nuyten MJ, Bartelink H. Bladder conservation in selected T1G3 and muscle-invasive T2-T3a bladder carcinoma using combination therapy of surgery and iridium-192 implantation. Br J Urol. 1994 Sep;74(3):322-7. doi: 10.1111/j.1464-410x.1994.tb16620.x. PMID 7953264
- [Result] Milowsky MI, Rumble RB, Booth CM, Gilligan T, Eapen LJ, Hauke RJ, Boumansour P, Lee CT. Guideline on Muscle-Invasive and Metastatic Bladder Cancer (European Association of Urology Guideline): American Society of Clinical Oncology Clinical Practice Guideline Endorsement. J Clin Oncol. 2016 Jun 1;34(16):1945-52. doi: 10.1200/JCO.2015.65.9797. Epub 2016 Mar 21. PMID 27001593
- [Result] Ploussard G, Daneshmand S, Efstathiou JA, Herr HW, James ND, Rodel CM, Shariat SF, Shipley WU, Sternberg CN, Thalmann GN, Kassouf W. Critical analysis of bladder sparing with trimodal therapy in muscle-invasive bladder cancer: a systematic review. Eur Urol. 2014 Jul;66(1):120-37. doi: 10.1016/j.eururo.2014.02.038. Epub 2014 Feb 26. PMID 24613684
- [Result] Rodel C, Grabenbauer GG, Kuhn R, Papadopoulos T, Dunst J, Meyer M, Schrott KM, Sauer R. Combined-modality treatment and selective organ preservation in invasive bladder cancer: long-term results. J Clin Oncol. 2002 Jul 15;20(14):3061-71. doi: 10.1200/JCO.2002.11.027. PMID 12118019
- [Result] Pieretti A, Krasnow R, Drumm M, Gusev A, Dahl DM, McGovern F, Blute ML, Shipley WU, Efstathiou JA, Feldman AS, Wszolek MF. Complications and Outcomes of Salvage Cystectomy after Trimodality Therapy. J Urol. 2021 Jul;206(1):29-36. doi: 10.1097/JU.0000000000001696. Epub 2021 Feb 22. PMID 33617327
- [Result] Herskind C, Bentzen SM, Overgaard J, Overgaard M, Bamberg M, Rodemann HP. Differentiation state of skin fibroblast cultures versus risk of subcutaneous fibrosis after radiotherapy. Radiother Oncol. 1998 Jun;47(3):263-9. doi: 10.1016/s0167-8140(98)00018-8. PMID 9681889